CLINICAL TRIAL: NCT01332942
Title: Randomized, Single-blind, Placebo-controlled, Combined Single / Multiple Dose Escalation, Group Comparison Study to Investigate Safety, Tolerability, Pharmacodynamic Effect and Pharmacokinetics of BAY 85-3934 in Patients With Renal Anemia Due to CKD (Stages 3 and 4)
Brief Title: Combined Single / Multiple Dose Escalation Study in Patients With Renal Anemia Due to CKD (Chronic Kidney Disease)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 14627; 2010-023585-50 (EudraCT Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Anemia
Keywords: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: BAY85-3934
- Molidustat (BAY85-3934) 5 mg (Experimental)
  Interventions: Drug: BAY85-3934
- Molidustat (BAY85-3934) 10 mg (Experimental)
  Interventions: Drug: BAY85-3934
- Molidustat (BAY85-3934) 25 mg (Experimental)
  Interventions: Drug: BAY85-3934
- Molidustat (BAY85-3934) 50 mg (Experimental)
  Interventions: Drug: BAY85-3934
- Molidustat (BAY85-3934) 75 mg (Experimental)
  Interventions: Drug: BAY85-3934

INTERVENTIONS:
Drug: BAY85-3934 — Subjects received an oral single dose of placebo tablet matched to the molidustat dose (BAY85-3934) on Day 1 followed by a washout day and once daily multipledose over 12 days (from Day 3 to Day 14).
  Arms: Placebo
Drug: BAY85-3934 — Subjects received an oral single dose of 5 mg of molidustat IR tablet on Day 1 followed by a washout day and once daily multiple-dose over 12 days (from Day 3 to Day 14).
  Arms: Molidustat (BAY85-3934) 5 mg
Drug: BAY85-3934 — Subjects received an oral single dose of 10 mg of molidustat ( 2x 5mg IR tablets) on Day 1 followed by a washout day and once daily multipledose over 12 days (from Day 3 to Day 14).
  Arms: Molidustat (BAY85-3934) 10 mg
Drug: BAY85-3934 — Subjects received an oral single dose of 25 mg of molidustat (1 x 20 mg IR tablet and 1 x 5 mg IR tablet) on Day 1 followed by a washout day and once daily multiple-dose over 12 days (from Day 3 to Day 14).
  Arms: Molidustat (BAY85-3934) 25 mg
Drug: BAY85-3934 — Subjects received an oral single dose of 50 mg) of molidustat (2 x 20 mg IR tablets and 2 x 5 mg IR tablets) on Day 1 followed by a washout day and once daily multiple-dose over 12 days (from Day 3 to Day 14).
  Arms: Molidustat (BAY85-3934) 50 mg
Drug: BAY85-3934 — Subjects received an oral single dose of 75 mg of molidustat (3 x 20 mg IR tablets and 3 x 5 mg IR tablets) on Day 1 followed by a washout day and once daily multiple-dose over 12 days (from Day 3 to Day 14).
  Arms: Molidustat (BAY85-3934) 75 mg

SUMMARY:
The drug that is under investigation during this study is BAY85-3934 which is intended to be used as a treatment for patients suffering from renal anemia due to chronic kidney disease (stage 3 and 4).

The purpose of this study is to provide safety and tolerability information on the drug. Other objectives of the study are to investigate the effect of the drug on the body (pharmacodynamics) as well as the absorption, breakdown, metabolism, distribution and excretion (pharmacokinetics) by measuring the concentration in blood and urine.

The study will be conducted in one study center in the United Kingdom and several centers in Germany. 84 (of which 36 are optional) patients who meet the inclusion criteria will participate in the study. BAY 85-3934 will be given following a combined single / multiple dose escalation design in seven (of which three are optional) dose steps.

ELIGIBILITY:
Inclusion Criteria:

The informed consent must be signed before any study specific tests or procedures are done

* Renal anemia due to CKD (stage 3 and 4) not on dialysis assessed by medical history and Creatine Clearance (CLCR) between 15 to 59 mL/min ± 10 % (ie CLCR between 13 - 65 mL/min) estimated at the pre-study visit from the creatinine concentration measured in serum (Modification of Diet in Renal Disease (MDRD) formula)
* Stable renal disease, ie without major changes in therapy within the last 6 weeks and not expected to begin dialysis within the study.
* Female subjects with no child-bearing potential (postmenopausal women with 12 month of spontaneous amenorrhea or with 6 month of spontaneous amenorrhea and serum FSH levels > 30 mIU/mL, women with 6 weeks post bilateral ovariectomy, woman with bilateral tubal ligation, and women with hysterectomy).
* Male subjects who agree to use two forms of effective contraception during the study and for 12 weeks after receiving the study drug. This must include a condom with spermicide gel for 21 days after drug administration.
* Male subjects who agree not to act as sperm donors for 12 weeks after dosing.
* Age: ≥ 18 and ≤ 85 years at the pre-study visit
* Body mass index (BMI): ≥ 18 and ≤ 35 kg / m2 at the pre-study visit
* Hemoglobin (Hb) of 8.0 - 12 g/dL (male) or 8.0 - 11.5 g/dL (female) at two consecutive measurements (1 measurement performed within 12 weeks to 2 days before the pre-study visit during routine diagnostics independently of the study and 1 measurement at the pre-study visit)
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Patients with impaired liver function (Child Pugh B and C based on medical history)
* Patients with hemolysis/hemolytic anemia or active bleeding/blood loss
* Major surgery or an intervention causing relevant blood loss or inflammation within the last 2 month
* Planned intervention or surgery during the study which might impact the study objectives.
* Febrile illness within 1 week before the first study drug administration or clinically significant infection.
* Patients with chronic inflammatory diseases (eg systemic lupus erythematosis, rheumatoid arthritis, Crohn´s disease) that could impact erythropoiesis or with persistent inflammatory activity (eg C-reactive protein (CRP) > 20mg/L)
* History of thrombotic or thromboembolic events (e.g. myocardial infarction, stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within the recent 6 months
* Proliferative choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy that required or is likely to require treatment (intraocular injections or laser photocoagulation) during the study.
* History of myelodysplastic syndrome, multiple myeloma, bone marrow fibrosis, or pure red cell aplasia.
* History of hemosiderosis or hemochromatosis.
* Patients with a history of malignant disease during the last 5 years
* Treatment with erythropoiesis stimulating agents (ESA) within the last 4 weeks before first intake of study drug
* Intravenous iron substitution 2 weeks before and during the treatment period with BAY 85-3934
* RBC transfusion during previous 8 weeks
* Use of products containing carnitine and/or anabolics
* Use of medicines or substances which oppose the study objectives or which might influence them within 14 days before the first study drug administration
* Significant uncorrected rhythm or conduction disturbances such as a second- or third-degree AV block without a cardiac pacemaker or episodes of sustained ventricular tachycardia
* Systolic blood pressure below 100 or above 160 mmHg at the pre-study visit
* Diastolic blood pressure below 50 or above 100 mmHg at the pre-study visit
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus antibodies (anti-HIV 1+2) at the pre-study visit
* Heart rate above 110 bpm
* Ferritin levels ≤ 30 ng/mL at the pre-study visit
* Transferrin-saturation < 15% at the pre-study visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Treatment-Emergent Adverse Events (TEAE) | From start of study drug administration until last follow-up visit (14 days after the last study drug administration)
  An adverse event (AE) was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important serious event. TEAEs were defined as AEs/SAEs that started or worsened after the study drug treatment.
Mean Change in Heart Rate Within 4 hours Post-dose | Within 4 hours from after administration of study drug on Day 1 and Day 14
  Heart rate was observed in all treatment groups in supine position.
Mean Change in Heart Rate Over 1 Minute for Doses 25, 50, 75 Milligrams | From start of study drug administration until 12 hours after the last study drug administration
  Heart rate was assessed over 1 minute from the Electrocardiogram (ECG) recording.
Mean Change in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Within 4 hours Post-dose | Within 4 hours post-dose at Day 1 and Day 14
  SBP, DBP was observed in all treatment groups in supine phase.
Number of Subjects with Clinically Relevant Abnormal Findings in the Electrocardiogram (ECG) | Day 1 and Day 14
  Electrocardiograms were recorded and analyzed by an electronic ECG reading system.
Number of Subjects with Clinically Relevant Laboratory Values | Day 1 and Day 14
  Laboratory parameters include hematology, coagulation, serum chemistry, urinalysis.
Maximum Observed Drug Concentration (Cmax) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  Cmax refers to the highest measured drug concentration after a single dose which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration Divided by Dose (Cmax/D) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  Cmax/D is defined as maximum observed drug concentration divided by dose. Cmax refers to the highest measured drug concentration after single dose which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  AUC is a measure of systemic drug exposure after single dose, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC is defined as area under concentration versus time curve from time 0 (pre-dose) to extrapolated infinite time. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Infinity Divided by Dose (AUC/D) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  AUC is a measure of systemic drug exposure after single dose, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC is defined as area under concentration versus time curve from time 0 (pre-dose) to extrapolated infinite time. AUC/D is defined as area under the concentration versus time curve from zero to infinity divided by dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration (Cmax,md) in Plasma of Molidustat and its Metabolite After Multiple Dose Administration of Molidustat | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  Cmax,md defined as maximum observed drug concentration after multiple dose. Cmax,md refers to the highest measured drug concentration in the dosing interval which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration in Plasma Divided by Dose (Cmax,md/D) of Molidustat and its Metabolite After Multiple Dose Administration of Molidustat | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  Cmax,md/D is defined as maximum observed drug concentration divided by dose after multiple dose administration. Cmax,md refers to the highest measured drug concentration within the dosing interval which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From 0 to 24 hour (AUC[0-24]md) in Plasma During any Dose Interval of Molidustat and its Metabolite After Multiple Dose of Molidustat | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  AUC(0-24)md is defined as area under the concentration versus time curve from 0 to 24 hour after multiple dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From 0 to 24 hour Divided by Dose (AUC[0-24] md/D) in Plasma During any Dose Interval of Molidustat and its Metabolite After Multiple Dose of Molidustat | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  AUC(0-24)md/D is defined as area under the concentration versus time curve from 0 to 24 hour divided by dose after multiple dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration in Plasma Divided by Dose per Kilogram Body Weight (Cmax,norm) of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Cmax,norm is defined as maximum observed drug concentration divided by dose per kilogram body weight. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Infinity in Plasma Divided by Dose per Kilogram Body Weight (AUCnorm) of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  AUC is a measure of systemic drug exposure after single dose, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUCnorm is defined as area under the concentration versus time curve from zero to infinity divided by dose per kilogram body weight. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to 24 hour (AUC[0-24]) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-24 hours post-dose
  AUC(0-24) is defined as area under the concentration versus time curve from zero to 24 hours after a single dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to the Last Data Point Above the Lower Limit of Quantification (AUC[0-tlast]) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  AUC is a measure of systemic drug exposure after single dose, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-tlast) is defined as AUC from time zero to the last data point above the lower limit of quantification. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Half Life Associated With the Terminal Slope (t1/2) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  Half life associated with terminal slope. It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase. It is expressed in hours and derived from the terminal slope of the concentration versus time curve. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time to Reach Maximum Drug Concentration (tmax) in Plasma of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content. Median and range were reported.
Mean Residence Time (MRT) of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  MRT is an average duration of the drug in the body, and is expressed in hours. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Apparent Oral Clearance (CL/F) of Molidustat and its Metabolite After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Apparent Volume of Distribution During Terminal Phase (Vz/F) After Single Dose of Molidustat | Single dose: 0-48 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the observed plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Amount Excreted into Urine (Aeur) of Molidustat and its Metabolite After Single Dose of Molidustat | Urine collection intervals: 0d00 - 0d12h, 0d12h - 1d00
  Aeur refers to the amount of molidustat excreted in urine.
Renal Body Clearance of Drug (CLR) of Molidustat and its Metabolite After Single Dose of Molidustat | Urine collection interval: 0d00 - 1d00
  Renal clearance describes the removal of drug from a volume of plasma in a given unit of time by the kidneys. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Concentration Divided by Dose per Kilogram Body Weight (Cmax,md,norm) in Plasma After Multiple Dose Administration During a Dosage Interval | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Cmax,md,norm is defined as maximum observed concentration during a given dosing interval divided by dose per kilogram body weight in plasma after multiple dose administration. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From 0 to 24 hour Divided by Dose per Kilogram Body Weight (AUC[0-24]md,norm) in Plasma After Multiple Dose Administration During a Dosage Interval | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-24) md,norm is defined as area under the concentration versus time curve from 0 to 24 hour divided by dose per kilogram body weight after multiple dose administration. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Half Life Associated With the Terminal Slope (t1/2,md) in Plasma of Molidustat and its Metabolite After Multiple Dose of Molidustat | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  Half life associated with terminal slope. It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase. It is expressed in hours and derived from the terminal slope of the concentration versus time curve. t1/2,md is defined as half life associated with the terminal slope after multiple dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time to Reach Maximum Drug Concentration (tmax,md) in Plasma of Molidustat and its Metabolite After Multiple Dose of Molidustat | Multiple dose: 0-24 hours post dose on Day 14 (13d)
  tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content. tmax,md is defined as time to reach maximum drug concentration after multiple dose. Median and range were reported.
Amount Excreted into Urine (Aeur,md)of Molidustat and its Metabolite After Multiple Dose of Molidustat | Urine collection interval: 13d00 - 14d00
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Renal Body Clearance (CLR,md) of Molidustat and its Metabolite After Multiple Dose of Molidustat | Urine collection interval: 13d00 - 14d00
  Renal clearance describes the removal of drug from a volume of plasma in a given unit of time by the kidneys. CLR,md is defined as renal body clearance of drug after multiple dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Accumulation Ratio of AUC in the Dosing Interval (RAAUC) of Molidustat | All samples from 0-24h on 0d and from 0-24h on 13d
  RAAUC was calculated by using formula AUC(0-24)[13day] / AUC(0-24)[0day].
Accumulation Ratio of Cmax (RACmax) of Molidustat | All samples from 0-24h on 0d and from 0-24h on 13d
  RACmax was calculated by using formula Cmax[13day] / Cmax[0day].
Linearity Factor of Pharmacokinetics After Repeated Administration of Identical Doses (RLin) of Molidustat | All samples from 0-24h on 0d and from 0-24h on 13d
  RLin was calculated by using formula AUC(0-24)[13day] / AUC[0day].
Erythropoietin Concentration: Area Under the Concentration Versus Time Curve From 0 to 24 hour (AUC[0-24]) Post-dose on Day 1 (0d) | Single dose: Pre-dose and 4, 8, 12 and 24 hours post-dose
  AUC(0-24) is defined as area under the concentration versus time curve from zero to 24 hours after a single dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Erythropoietin Concentration: Area Under the Concentration Versus Time Curve From 0 to 24 hour (AUC[0-24]md) in Plasma After Multiple Dose on Day 14 (13d) | Multiple dose: Pre-dose and 4, 8, 12 and 24 hours post-dose on 13day
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Erythropoietin Concentration: Maximum Observed Drug Concentration in Plasma (Cmax[0-24]) After Single Dose of Molidustat on Day 1 (0d) | Single dose: Pre-dose and 4, 8, 12, 24 hours post-dose
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Erythropoietin Concentration: Maximum Observed Drug Concentration in Plasma (Cmax [0-24]md) Within 0-24 hours Post Dose on Day 14 (13d) | Multiple dose: Pre-dose and 4, 8, 12 and 24 hours post-dose on 13day
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Pharmacodynamic Parameter: Maximum Observed Drug Concentration in Plasma (Cmax) of Reticulocytes (Absolute) Within Day 1 (0d) - Day 14 (13d) | Day 1 to Day 14
Pharmacodynamic Parameter: Maximum Observed Drug Concentration in Plasma (Cmax) of Reticulocytes ( Ratio-to-Baseline-Adjusted) Within Day 1(0d) - Day 14 (13d) | Day 1 to Day 14
Pharmacodynamic Parameter: Maximum Observed Drug Concentration in Plasma (Cmax) of Hemoglobin (Absolute) Within Day 1 (0d) - Day 14 (13d) | Day 1 to Day 14
Pharmacodynamic Parameter: Maximum Observed Drug Concentration in Plasma (Cmax) of Hemoglobin ( Ratio-to-Baseline-Adjusted) Within Day 1 (0d) - Day | Day 1 to Day 14
Pharmacodynamic Parameter: Maximum Observed Drug Concentration in Plasma (Cmax) of Hematocrit (Absolute) Within Day 1 (0d) - Day 14(13d) | Day 1 to Day 14
Pharmacodynamic Parameter: Maximum Observed Drug Concentration in Plasma (Cmax) of Hematocrit (Ratio-to-Baseline-Adjusted) Within Day 1( 0d) - Day 14 (13d) | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- Germany (8):
  - München, Bavaria
  - Hamburg, Hamburg
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Kiel, Schleswig-Holstein
  - Berlin, State of Berlin
  - Wuppertal
- London, London, United Kingdom

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/